CLINICAL TRIAL: NCT05651958
Title: Effects of Pranayama Breathing Technique on Dyspnea, Exercise Tolerance and Quality of Life in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Effects of Pranayama Breathing Technique in Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/22/0351 Amina Muqaddas
Record Dates: First submitted 2022-12-06; First posted 2022-12-15 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Pranayama; COPD; Dyspnea; Exercise tolerance
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea | interventions — Nebulizers and Vaporizers

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pranayma Breathing Technique (Experimental): Pranayma Breathing Technique protocol includes 15 breaths in the morning and 15 breaths in evening for atleast weeks.
  Interventions: Other: Breathing Technique
- Conventional Treatment (Active Comparator): Long-acting beta-2 agonist, nebulizers and long acting anti-mucosic drugs.
  Interventions: Other: Nebulizer

INTERVENTIONS:
Other: Nebulizer — Active Comparator: Nebulization every 3 days with the other medicine to the active comparator.
  Arms: Conventional Treatment
Other: Breathing Technique — 15 repeatations of Breathing in morning and evening
  Arms: Pranayma Breathing Technique

SUMMARY:
It will be randomized controlled trial. The research will be conducted at Bahawal Victoria hospital Bahawalpur and civil hospital Bahawalpur. We take 60 patients (Epitool), Patients will be allocated randomly in two groups. Group A will get conventional medical treatment and Group B will get both conventional medical treatment and pranayama breathing exercise. Both gender of age group 30 to 55, Patient with diagnosed Chronic obstructive pulmonary disease ,Moderate to severe Chronic obstructive pulmonary disease with productive cough, Shortness of breathe and no surgical procedure performed will be included in this study. And patients of lung surgery, lung cancer, above 70 years age, with open wound, cardiovascular issues, and neurological issues will be excluded. Yoga exercise pranayama, 6 min walk test, IPAQ- quality of life and VSAQ-exercise capacity will be used as tools. Data will be analyzed on SPSS 21.

DETAILED DESCRIPTION:
It will be randomized controlled trial. After approval of synopsis the research will be conducted at Bahawal Victoria hospital Bahawalpur and Sadiq abbasi hospital Bahawalpur. Written informed consent will be obtained. We take 60 patients (Epitool), Patients will be allocated randomly in two groups. Group A and group B. Group A will get conventional medical treatment and Group B will get both conventional medical treatment and pranayama breathing exercise. Both gender of age group 30 to 55, Patient with diagnosed COPD, Moderate to severe COPD with productive cough, SOB and no surgical procedure performed will be included in this study. And patients of lung surgery, lung cancer, above 70 years age, with open wound, cardiovascular issues, and neurological issues will be excluded. Yoga exercise pranayama, 6 min walk test, IPAQ- quality of life and VSAQ-exercise capacity will be used as tools. Data will be analyzed on SPSS 21.

ELIGIBILITY:
Inclusion Criteria:

* Both gender of age group 30 to 55

  * Patient with diagnosed COPD.
  * Moderate to severe COPD.
  * Patient with productive cough and SOB.
  * No surgical procedure perform.

Exclusion Criteria:

* Patient of lung surgery

  * Lung cancer patient
  * Patient above 70 years age.
  * Patient with open wound.
  * Patient with cardiovascular issues

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
6 min walk test. | Six Weeks
  The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
IPAQ- quality of life | Six Weeks
  The International Physical Activity Questionnaire (IPAQ) will be used to evaluate the current physical activity level of the participants.
VSAQ-exercise capacity | Six Weeks
  The VSAQ, capturing patient-reported outcome measures, is an efficient and quantifiable measure of exercise capacity that can be readily employed in clinical services particularly where patients have normal to high exercise tolerance

CONTACTS AND LOCATIONS:
Overall Officials: madiha younas, MS, Principal Investigator — riphah internationl university
Locations (1):
- Bahawal Victoria Hospital and Civil Hospital, Chak Four Hundred Fifty-four, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No